CLINICAL TRIAL: NCT06589778
Title: Safety, Tolerability, and Efficacy of SHR-A2102 in Combination With Adebrelimab, With SHR-8068, in Subjects With Locally Advanced or Metastatic Non-Small Cell Lung Cancer: A Phase IB/II Open-Label, Multicenter Clinical Study
Brief Title: A Study of SHR-A2102 in Combination With Adebrelimab and SHR-8068 in Subjects With Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A2102-206
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-09

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-A2102 in Combination with Adebrelimab and SHR-8068 (Experimental)
  Interventions: Drug: SHR-A2102; Drug: Adebelimab (SHR-1316); Drug: SHR-8068

INTERVENTIONS:
Drug: SHR-A2102 — SHR-A2102: injection, 80mg/ bottle, intravenous drip
Drug: Adebelimab (SHR-1316) — Adebelimab (SHR-1316): injection, 600mg(12mL)/ bottle, intravenous drip
Drug: SHR-8068 — SHR-8068: injection, 50mg（10mL）/ bottle, intravenous drip

SUMMARY:
This study is a multicenter, open-label, dose-finding/efficacy-expanding Phase IB/II clinical trial to evaluate SHR-A2102 in combination with adebelimab in combination with SHR-8068 in patients with locally advanced or metastatic non-small cell lung cancer. The study consists of two phases: Phase IB to explore the safety/tolerability of SHR-A2102 in combination with adebelimab in combination with SHR-8068 in patients with locally advanced or metastatic non-small cell lung cancer; Phase II: To explore the efficacy of SHR-A2102 in combination with adebelimab in combination with SHR-8068 in patients with locally advanced or metastatic non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects are able to give voluntary informed consent, understand the study and are willing to follow and complete all the test procedures.
2. Age 18~70 years old.
3. Pathologically confirmed unresectable locally advanced/metastatic non-small cell lung cancer.
4. At least one measurable lesion per RECIST v1.1 criteria.
5. ECOG PS score: 0-1.

Exclusion Criteria:

1. Active or symptomatic brain metastases.
2. Previous diagnosis of any other malignancy.
3. Clinically symptomatic moderate to severe ascites; Uncontrollable or moderate or above pleural effusion, pericardial effusion.
4. Received anti-tumor therapy 4 weeks prior to initiation of study treatment.
5. Uncontrolled tumor-related pain.
6. Subjects with severe cardiovascular and cerebrovascular diseases.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-09-27 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Determination of Recommended Phase II dose (RP2D) | From first dose of study treatment until the end of Cycle 1（up to 21 days）
Objective Response Rate (ORR) | From time of first dose of SHR-A2102 or Adebrelimab or SHR-8068 until the date of objective disease progression or death (up to 12 months)
  The percentage of participants with a confirmed CR or PR according to RECIST v1.1 criteria.
Incidence and severity of AEs | The observation period ended at the end of the 21-day period after the first dose of SHR-A2102 or Adebrelimab or SHR-8068 (up to 21 days)

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | From time of first dose of SHR-A2102 or Adebrelimab or SHR-8068 until the date of objective disease progression or death (up to 12 months)
  The percentage of participants who have a best objective response of confirmed CR or PR or who have SD after start of treatment.
Duration of Response (DoR) | From time of first dose of objective disease progression until the date of objective disease progression or death (up to 12 months)]
  The time from the date of first response until date of disease progression or death in the absence of disease progression.
Progression free Survival (PFS) | From time of first dose of objective disease progression until the date of objective disease progression or death (up to 12 months)
  Progression-free survival is defined as the time from the start of treatment until the date of objective disease progression or death.
Overall Survival (OS) | From time of first dose of objective disease progression until the date of death (up to 24 months)
  The time until death due to any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided